CLINICAL TRIAL: NCT02654301
Title: Beneficial Effect of Xylose Consumption on Postprandial Hyperglycemia in Subjects With Normal Glucose Level and Impaired Fasting Glucose
Brief Title: Beneficial Effect of Xylose Consumption on Postprandial Hyperglycemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Jong Ho Lee, Department of Food and Nutrition, Yonsei University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Xylose_2015
Record Dates: First submitted 2015-08-26; First posted 2016-01-13 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2015-08

CONDITIONS: Postprandial Hyperglycemia
Keywords: Xylose; prediabetes; postprandial hyperglycemia; glucose
MeSH Terms: conditions — Hyperglycemia; Prediabetic State

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control group (Placebo Comparator): sucrose drink (Control, sucrose 50g + deionized water 100g)
  Interventions: Dietary Supplement: Control
- 5 g xylose group (Active Comparator): 5 g xylose (Test 1, sucrose : xylose = 10:1),
  Interventions: Dietary Supplement: Test 1
- 3.33 g xylose group (Active Comparator): 3.33 g xylose (Test 2, sucrose : xylose = 15:1)
  Interventions: Dietary Supplement: Test 2
- 2.5 g xylose group (Active Comparator): 2.5 g xylose (Test 3, sucrose : xylose = 20:1)
  Interventions: Dietary Supplement: Test 3

INTERVENTIONS:
Dietary Supplement: Test 1 — sucrose : xylose = 10:1, sucrose 50 g + xylose 5 g + deionized water 95 g
  Arms: 5 g xylose group
Dietary Supplement: Test 2 — sucrose : xylose = 15:1, sucrose 50 g + xylose 3.33 g + deionized water 96.67 g
  Arms: 3.33 g xylose group
Dietary Supplement: Test 3 — sucrose : xylose = 20:1, sucrose 50 g + xylose 2.5 g + deionized water 97.5 g
  Arms: 2.5 g xylose group
Dietary Supplement: Control — sucrose 50 g + deionized water 100 g
  Arms: Control group

SUMMARY:
The present study determined the effect of Xylose consumption on postprandial hyperglycemia in normal (n=25) and hyperglycemic subjects (n=50).

DETAILED DESCRIPTION:
In this double-blind crossover designed study, Participants were randomly assigned to consume a sucrose drink (Control, sucrose 50g + deionized water 100g) or a sucrose drink additionally containing 5 g (Test 1, sucrose : xylose = 10:1), 3.33 g (Test 2, sucrose : xylose = 15:1) or 2.5 g (Test 3, sucrose : xylose = 20:1) of D-xylose with a week interval.

ELIGIBILITY:
Inclusion Criteria:

1) healthy subject or Impaired fasting glucose (fasting serum glucose between 100 and 125 mg/dL)

Exclusion Criteria:

1. history of taking an insulin-injection or oral hypoglycemic agents
2. evidence of alcohol abuse or alcoholism
3. pregnancy or breast feeding
4. chronic gastrointestinal disorder
5. seriously abnormal liver or renal function
6. an occupation at risk of death when hypoglycemia occurs

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-06; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change of serum glucose levels | a week interval

SECONDARY OUTCOMES:
Change of serum insulin levels | a week interval
Change of serum C-peptide levels | a week interval

CONTACTS AND LOCATIONS:
Overall Officials: Jong Ho Lee, Ph.D, Principal Investigator — Laboratory of clinical nutrigenetics/nutrigenomics, Yonsei University

REFERENCES:
- [Derived] Jun YJ, Lee J, Hwang S, Kwak JH, Ahn HY, Bak YK, Koh J, Lee JH. Beneficial effect of xylose consumption on postprandial hyperglycemia in Korean: a randomized double-blind, crossover design. Trials. 2016 Mar 15;17(1):139. doi: 10.1186/s13063-016-1261-0. PMID 26979433